CLINICAL TRIAL: NCT06752993
Title: Effects of Expiratory Muscle Strength Training on Cobb Angle, Respiratory Muscle Strength, Core Stabilization, Functional Exercise Capacity and Quality of Life in Adolescent Idiopathic Scoliosis
Brief Title: Effects of Expiratory Muscle Strength Training in Adolescent Idiopathic Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Associate Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02112001
Record Dates: First submitted 2024-12-06; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Scoliosis; Adolescence
Keywords: Adolescent idiopathic scoliosis; Expiratory muscle strength training; Cobb angle; Core stability; Functional exercise capacity; Respiratory muscle stregth
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Muscle Strength Training Group (Active Comparator): The treatment group will receive expiratory muscle strength training (EMST) at 50% maximal expiratory mouth pressure (PEmax) by using EMST-150 device and training load were adjusted to maintain 50% of the PEmax weekly. The PEmax will measured at supervised sessions each week and 50% of the measured value will determined as the new training work load.
  Interventions: Device: Expiratory Muscle Strength Training (EMST-150)
- Sham Group (Sham Comparator): The control group will receive expiratory muscle strength training (EMST) without physiological load by using expiratory muscle strength training device.
  Interventions: Device: Sham Training

INTERVENTIONS:
Device: Expiratory Muscle Strength Training (EMST-150) — Training is going to perform by using a pressure treshold-loading device (EMST-150, Aspire Products, LLC, Gainesville, FL) used to exhale against a same-pressure load every exhalation for strengthening primarily the core muscles. The device pressure is adjusted according to PEmax and reliability/reproducibility has been demonstrated.
  Arms: Expiratory Muscle Strength Training Group
Device: Sham Training — Training is going to perform by using a pressure treshold-loading device (EMST-150, Aspire Products, LLC, Gainesville, FL) without physiological load. The sham device closely resembled the EMST device, with the only difference being that the pressure release valve was rendered nonfunctional by removing the spring. As a result, it exerted minimal to no physiological load on the targeted muscles.
  Arms: Sham Group

SUMMARY:
Adolescent idiopathic scoliosis result in deterioration of core muscles and respiratory system. Core muscles provide trunk stabilization as well as responsible for respiratory system. Especially tr. abdominis, rectus abdominis, external oblic and internal oblic muscle, which are core muscles, highly active during forced expiration while diaphragm muscle also active during inspiration. Thus, expiratory muscle strength training has effect not only respiratory muscle strength but also trunk stabilization. While, effects of expiratory muscle strength training in adolesecent idiopathic scoliosis is a topic that needs to be investigated, this topic has not been investigated until today. Hence, this current study aimed to investigate the effects of expiratory muscle strength training on cobb angle, respiratory muscle strength, core stabilization, functional exercise capacity and quality of life.

DETAILED DESCRIPTION:
A convenience of children with adolescent idiopathic scoliosis, 10-19 years, is going to recruited from Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. Patients will randomly allocate to either a treatment group or control group. The treatments group will receive expiratory muscle strength training at 50% maximal expiratory presssure while, the control group will receive sham expiratory muscle strength training without physiological load. Groups are going to train for a total of 25 breathe/day, 5 days/week, for 6 weeks. Before and after treatment, all of patients progression of scoliosis will be evaluated by calculating cobb angle, respiratory muscle strength using with electronic mouth pressure device, core stability using with Mc-Gill endurance test and the stabilizer biofeedback unit, functional exercise capacity using with six minute walk test (6MWT) and six minute pegboard and ring test (6MPBRT), quality of life using with scoliosis research society -22 questionnare (SRS-22) and daily living activity of upper extremity using with quick-DASH questionnare.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with idiopathic scoliosis,
* aged between 10 and 19 years,
* with a Cobb angle ranging from 10 to 45 degrees.

Exclusion Criteria:

* Individuals who have undergone spinal surgery,
* who have received conservative or surgical treatment for scoliosis,
* individuals with neurological, neuromuscular, systemic, rheumatological, or musculoskeletal disorders, or conditions affecting balance and walking,
* individuals with a history of cardiac or pulmonary diseases that could affect respiratory function and exercise capacity.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-04 (Estimated); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle | 6 Weeks
  This is the gold standard method used to assess the lateral curvature of the spine. In this method, participants' anteroposterior radiographic images will be captured while they are in a standing position. The angle between a line drawn parallel to the upper edge of the highest vertebra involved in the scoliosis curve and a line drawn parallel to the lower edge of the lowest vertebra involved will be measured on the radiographic image. These measurements will be performed by an experienced orthopedic physician

SECONDARY OUTCOMES:
Respiratory Muscle Strength | 6 Weeks
  The measurement of maximal inspiratory pressures (MIP) and maximal expiratory pressures (MEP), which are voluntarily assessed to evaluate the participants' respiratory muscle strength, will be conducted using an electronic and portable mouth pressure measurement device (Micro Medical MicroRM, UK) in accordance with ATS/ERS criteria.
McGill Endurance Test | 6 Weeks
  The participants' core stabilization will be assessed using the McGill Endurance Test.
'6 Minute Pegboard and Ring' Test | 6 Weeks
  To assess the functional exercise capacity of the participants, the 'Pegboard and Ring' test will be performed for the upper extremities.
Scoliosis Research Society 22 Patient Questionnaire | 6 Weeks
  The participants' quality of life will be assessed using the scoliosis research society 22 patient questionnaire. This questionnaire consists of 22 items and each item is scored between 0-5 point. While, the maximum score that obtained from the questionnaire is 110 point, the minimum score is 0 point. An increase scores on this questionnaire mean that quality of life has improved.
Quick Disabilities of the Arm, Shoulder and Hand Questionnaire | 6 Weeks
  The functional impairments of the upper extremities in the participants' activities of daily living will be assessed using the quick disabilities of the arm, shoulder, and hand questionnaire. This questionnaire consists of 11 items and each item is scored between 1-5 point. While, the maximum score that obtained from the questionnaire is 55 point, the minimum score is 11 point. An increase scores on this questionnaire mean that upper extremities in the participants' activities of daily living have worsened.
The Stabilizer Pressure Biofeedback Unit | 6 Weeks
  To assess the deep core muscle stabilization of the participants, the stabilizer pressure biofeedback unit will be performed.
6 Minute Walk Test | 6 Weeks
  To evaluate functional exercise capacity of the participants, the '6-Minute Walk test will be conducted for the lower extremities

CONTACTS AND LOCATIONS:
Overall Officials: Muserrefe Nur Keles, PhD, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No